CLINICAL TRIAL: NCT04437693
Title: Post Exposure Prophylaxis (PEP) in Healthcare Workers Exposed to COVID-19 Patients: A Double-blind Randomized Clinical Trial
Brief Title: Post Exposure Prophylaxis in Healthcare Workers Exposed to COVID-19 Patients
Acronym: HCQ-COVID19
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MRC-02-20-442
Record Dates: First submitted 2020-06-17; First posted 2020-06-18 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-06

CONDITIONS: COVID 19
Keywords: Hydroxychloroquine; Coronavirus Disease 2019; Post Exposure Prophylaxis; Center for Disease Control and Prevention; Coded Record Form
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: An interventional, double-blind, placebo-controlled randomized trial
Who Masked: Participant
Masking Description: The process of keeping the study group assignment hidden after allocation will be used where the investigator and participants will be unaware of the drug.A double blind randomized clinical trial has been proposed having 250 subjects in each arm. 500 subjects will be selected using randomly permuted blocks of 2,4, and 8 for the random process to allocate subjects into the two groups equally by using computer software.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydroxychloroquine (Experimental): 400mg twice a day on day 1 followed by 400 mg weekly for 7 weeks.
  Interventions: Drug: Hydroxychloroquine
- Placebo (Placebo Comparator): 2 tablets (Placebo White tablets) twice daily on day 1 followed by 2 tablets weekly for 7 weeks
  Interventions: Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Hydroxychloroquine — The treatment group that will receive Hydroxychloroquine (HCQ) 400mg twice a day on day 1 followed by 400 mg weekly for 7 weeks
  Other Names: Placebo

SUMMARY:
More cases of COVID-19 pandemic are being reported daily around the world. It is highly infectious and, over 7 million people have been infected and more than 400,000 people have died globally till this date. Countries around the world are struggling to avoid the spread of this pandemic.

Center for Disease Control and Prevention (CDC) confirmed that there are no approved drugs for COVID-19 treatment. Researchers around the globe, however, are researching different medications for COVID-19 patients, including the drug Hydroxychloroquine (HCQ), which is mainly used for Rheumatoid Arthritis and Malaria. Not enough data was obtained yet to know how well all of these medications are functioning. Therefore, aim to perform a randomized placebo-controlled trial to assess the impact of these medications on COVID -19 healthcare workers exposed while treating COVID 19 patients in Qatar to avoid causality and comorbidities in healthcare workers.

It is considered as a weak base. Many viruses enter the host cells via endocytosis, as a result of which they are initially taken up into an intracellular compartment that is "typically fairly acidic" whereas; Hydroxychloroquine would alter the acidity of this compartment, which can interfere with the ability of viruses to escape into the host cell and start replicating. Another hypothesis on the rationale of the Antiviral activity of HCQ, is that HCQ may also alter the ability of the virus to bind to the outside of a host cell in the first place.

An interventional, double-blind, placebo-controlled randomized trial that will include participants who will be healthcare workers at risks of exposure to COVID-19 while managing patients with confirmed infection.

Study will compare the safety, efficacy and effectiveness of Post Exposure Prophylaxis (PEP) use of HCQ in healthcare workers at risk of exposure to COVID-19 patients, in comparison to Placebo in Qatar.

DETAILED DESCRIPTION:
More cases of COVID-19 pandemic are being reported daily around the world. It is highly infectious and, over 7 million people have been infected and more than 400,000 people have died globally till this date. Countries around the world are struggling to avoid the spread of this pandemic. The most common symptoms of coronavirus disease are fever, fatigue, and dry cough. Most people (approximately 80 percent) recover from the disease without special care. The disease can be serious, and even fatal. Older people, and people with other medical conditions (such as asthma, diabetes, or heart disease), maybe more vulnerable to becoming severely ill. As the COVID-19 pandemic continues to affect communities throughout the world, the search for effective drugs remains a priority. Scientists across the globe are working to produce a vaccine, but unlikely to be available before 2021. Meanwhile, a growing number of countries have taken a series of systematic measures to curb coronavirus spread, including national lockdowns, meeting bans, school closings, closures of restaurants, bars, sports clubs etc

Researchers used to evaluate the invitro effectiveness of several potential COVID-19 treatments, including chloroquine (CQ) and redmeveir (RDV). The findings were found encouraging as 90 percent of the virus was inhibited by a low concentration of CQ and the results for RDV were even better-with an even lower concentration of this drug, achieving a virus inhibition of 90 percent. However, unless clinically verified, it cannot confirm these drugs for the treatment of COVID-19 patients. It is not known how well these medications function in people who are infected with COVID-19 and is still being studied. The first patient reported to be infected with COVID -19 in the U.S. was treated with RDV. The treatment started on the 7th day of hospitalization and on the 11th day after his symptoms were first identified. He started showing signs of progress on the very next day, presumably due to treatment with RDV. Further data, however, is required to confirm the effect of this treatment.

Researchers in France have also been studying the effectiveness of hydroxychloroquine (HCQ) in a single-arm regimen to treat people with COVID-19. HCQ (and, in some cases, also antibiotic azithromycin) has been used in this study to treat individuals with the COVID-19 virus in one setting. Investigators measured the amount of virus in swabs taken from these individuals and from a group of individuals who did not receive HCQ. A larger decrease in the volume of the virus from the individuals receiving HCQ occurred on a span of six days. However, the groups were not randomized. Individuals who did not receive HCQ were at various medical facilities and not necessarily like the individuals in the HCQ group. The results are intriguing. But it's important to note that scientists have expressed concerns about this study. Indeed, after the publication of these findings, a statement has been released in the journal that it did not meet the "expected standard" of research (6).

Moreover, these two drugs HCQ and RDV were designed primarily to fight other diseases and not COVID-19. Few data are available indicating that either could have some interest in the treatment of the disease, but its complete effect on COVID-19 patients is not known. One reason why researchers are interested in this drug is the HCQ's ability to modulate the inflammatory response. Inflammation is the natural reaction of the body to bacteria, viruses, or other substances that attack it. Our immune system usually attacks and actively kills infected cells or foreign bodies. But this response may often fail to function properly particularly in autoimmune disorders where the body is mistakenly attacking itself. HCQ has subtle effects on a wide variety of immune cells, and it may be that one of these effects helps stimulate the body's ability to fight off Covid-19. The inflammatory response in COVID-19 can be so strong that it causes serious damage to the lungs, that is why patients with severe infections need ventilators

Another hypothesis on the rationale of the Antiviral activity of HCQ, is that HCQ may also alter the ability of the virus to bind to the outside of a host cell in the first place.

The gold standard of a drug trial is a placebo-controlled, randomized, double-blind study. One group of participants should receive the investigational drug and another group should receive a placebo. The individuals in each arm of the study should be randomized; the demographics of both groups should be similar. Finally, the participants should not know if they are receiving the investigational drug or a placebo and the healthcare workers should not know what they are administering. Only under these conditions, It can conclusively determine the safety and efficacy of a potential treatment.

Center for Disease Control and Prevention (CDC) confirmed that there are no approved drugs for COVID-19 treatment. Researchers around the globe, however, are researching different medications for COVID-19 patients, including the drug Hydroxychloroquine, which is mainly used for the treatment of Rheumatoid Arthritis and Malaria. Not enough data was obtained yet to know how well all of these medications are functioning. Therefore, aim to perform a randomized placebo-controlled trial to assess the impact of these medications on healthcare workers who exposed for the treatment of COVID -19 patients in Qatar.

Rational to conduct a clinical trial on HCQ: It is considered as a weak base. Many viruses enter the host cells via endocytosis, as a result of which they are initially taken up into an intracellular compartment that is "typically fairly acidic" whereas; Hydroxychloroquine would alter the acidity of this compartment, which can interfere with the ability of viruses to escape into the host cell and start replicating. Another hypothesis on the rationale of the Antiviral activity of HCQ, is that HCQ may also alter the ability of the virus to bind to the outside of a host cell in the first place.

Hypothesis:

HCQ will be more safe and effective in comparison to placebo in the prevention of COVID 19 cases, in healthcare workers exposed to COVID 19 patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older, all healthcare workers in direct contact with COVID-19 patients (ex: physicians, nurses, pharmacists, etc.), the ability to swallow Oral medications, without any GI abnormalities that may affect absorption. Who agree to participate in the trial.

Exclusion Criteria:

* Allergy to HCQ.
* Pregnancy or breastfeeding.
* Known history of Retinal disease not related to Macular degeneration, or preexisting eye retinopathy.
* Having a prior history of blood disorders such as aplastic anemia, agranulocytosis, leukopenia, or thrombocytopenia.
* Having a prior history of glucose-6-phosphate dehydrogenase (G-6-PD) deficiency.
* Having dermatitis, psoriasis, or porphyria.
* History of lung disease or Pneumonia not related to COVID-19.
* Taking CYP450 enzyme-inducing medications within 4 weeks of the start of taking HCQ (Ex: Phenytoin, Carbamazepine, Phenobarbital, Primidone or Oxcarbazepine.
* Currently taking QT-prolonging medications, which may include Antiarrhythmics, Quinolones, Macrolides, select Antipsychotics and Antidepressants.
* Team members planning to have major abdominal, thoracic, spine or CNS surgery during the protocol period

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-08-31 (Estimated); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevention of SARS-CoV-2 infection | 7 Months
  Prevention of SARS-CoV-2 infection as determined by negative RT-PCR of the participants in the treatment group through swabbing that will be conducted on a weekly basis (Swabbing will be conducted at baseline and weekly through the end of the treatment period
Presence of any adverse effects related to HCQ | 7 months
  To find out the adverse effects related to HCQ such as : skin rashes, especially those made worse by sunlight, feeling sick (nausea) or indigestion, diarrhea, headaches, bleaching of the hair or mild hair loss, tinnitus (ringing in the ears) visual problem
Incidence of COVID-19 related symptoms | 7 weeks
  Incidence of COVID-19 related symptoms, that may include: Temperature over 37.8 degrees Celsius, Shortness of Breath, Cough.

CONTACTS AND LOCATIONS:
Overall Officials: Nasser Al Ansari, FRCPath, Principal Investigator — Hamad Medical Corporation (HMC)

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: One year
Access Criteria: 2021 to 2025

REFERENCES:
- Available data/document: Clinical Study Report — https://www.worldometers.info/coronavirus/ — https://www.worldometers.info/coronavirus/
- Available data/document: Clinical Study Report — https://www.who.int/docs/default-source/coronaviruse/who-china-joint-mission-on-covid-19-final-report.pdf — https://www.who.int/docs/default-source/coronaviruse/who-china-joint-mission-on-covid-19-final-report.pdf